CLINICAL TRIAL: NCT06997328
Title: '5 Rs to Rescue' A Cluster Trial With an Embedded Process Evaluation
Status: Recruiting | Type: Observational
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Bruce Biccard, Co-Principal Investigator, University of Cape Town
Other Study IDs: '5 Rs to Rescue'
Record Dates: First submitted 2024-08-21; First posted 2025-05-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-05

CONDITIONS: Surgery; Failure to Rescue
Keywords: Quality improvement; Postoperative Mortality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High-risk surgical patients: High-risk patients (ASOS Surgical Risk Calculator Score >10) having surgery, defined as ≥7 high risk patients having surgery per week.
  Interventions: Other: Implementation of the '5 Rs to Rescue'

INTERVENTIONS:
Other: Implementation of the '5 Rs to Rescue' — Quality improvement intervention increases surveillance for patients at risk of 'failure to rescue' after surgery

SUMMARY:
'Failure to rescue' describes the preventable death of a patient following the absence of timely identification and treatment of a complication after surgery. The absence of systems contributes to the higher mortality post-surgery in Africa compared to high-income countries. To mitigate this, a complex quality improvement (QI) intervention has been designed focusing on improving five main areas of patient management following surgery termed as '5 Rs to Rescue'. The study will take place in 20 centers in 4 countries - Ethiopia, South Africa, Tanzania, and Uganda. This a multi-center, mixed methods, cluster trial with a baseline assessment to evaluate the efficacy of the QI intervention. To study is aimed to evaluate whether implementation of the '5 Rs to Rescue' quality improvement intervention increases surveillance for patients at risk of 'failure to rescue' after surgery in hospitals in Africa.

The '5 Rs to Rescue' includes:

1. Risk assessment using the ASOS risk score for all surgical patients,
2. Recognition of patient deterioration by regular, protocolized vital signs monitoring plus use of an Early Warning Score (EWS) system. 3. Response to deterioration by protocolized escalation based upon EWS plus protocolized care pathways for common complications (hypoxia, hypovolemia, sepsis). 4. Reassessment following deterioration by protocolized re-assessment based upon EWS, and 5. Reflection on care provided following a patient's deterioration or death using a structured review tool at regular reflection meetings.

DETAILED DESCRIPTION:
INTRODUCTION 'Failure to rescue' describes the preventable death of a patient following a complication after surgery. Patients who develop complications after surgery, such as haemorrhage or infection, begin to deteriorate physiologically and become acutely unwell. This is usually identified by careful monitoring of the patient's basic 'vital signs' which include pulse rate, respiratory rate, oxygen saturation, blood pressure and consciousness level. However, if physiological deterioration is not identified and treated in a timely manner, it will progress and lead to organ dysfunction and then organ failure. This will ultimately lead to cardio-respiratory arrest and the death of the patient. 'Failure to rescue' can be used as a key concept in delivering safe and effective perioperative care as well as a healthcare quality metric in general. The first African Surgical Outcomes Study (ASOS-1) showed that 'failure to rescue' is the mode of death in 19 out of 20 deaths following surgery across Africa. Hospitals in high-income countries use early warning systems to monitor patients after surgery and trigger the escalation of care for patients who are critically ill to ensure prompt treatment. However, these systems do not exist in many resource-poor African hospitals where nurse: patient ratios can be as high as 1:35 and limit capacity-to-rescue within the system. Furthermore, in many African hospitals early warning systems are not used to monitor patients following surgery. These factors contribute to the higher mortality post-surgery in Africa compared to high-income countries. As patient outcomes tend to improve when enhanced monitoring increases the identification and treatment of critically ill patients, the study has co-produced a complex intervention with healthcare staff, community engagement and involvement (CEI) partners, and the Institute for Health Improvement (IHI) across four African countries (Ethiopia, South Africa, Tanzania and Uganda) to improve the capacity-to-rescue. This is a multi-centre, cluster trial with a baseline assessment to evaluate the efficacy of the '5 Rs to Rescue' quality improvement intervention using a mixed-methods process evaluation of the trial intervention. The intervention focuses on improving five main areas of patient management following surgery: 1) Risk assessment, 2) Recognition of patient deterioration, 3) Response to patient deterioration, 4) Reassessment following intervention to manage deterioration, and 5) Reflection on care provided following a patient's death. The complex quality improvement (QI) intervention is known as '5 Rs to Rescue'. Ultimately, the researchers intend to conduct a large international cluster randomised trial of the '5 Rs to Rescue' intervention comparing patient important outcomes for patients undergoing major surgery between intervention and usual care hospitals. The study hopes to demonstrate that the intervention can decrease 'failure to rescue' in Africa, and improve postoperative survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older undergoing any surgery, who receive postoperative care on a participating ward

Exclusion Criteria:

* Patients who opt out of trial participation.
* Patients receiving end of life care.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical wards of participating hospitals in four African countries (Ethiopia, South Africa, Tanzania, Uganda).
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Report site specific interventions and findings that explain how and why the 5R's to Rescue Quality Improvement Programme was effective or not in reducing in-hospital death after surgery. | 72 hours after surgery
  The complex QI intervention is known as '5 Rs to Rescue'. Ultimately, the study intends to conduct a large international cluster randomised trial of the '5 Rs to Rescue' intervention comparing patient important outcomes for patients undergoing major surgery between intervention and usual care hospitals. The study is aiming to demonstrate that the '5 Rs to Rescue' intervention can decrease 'failure to rescue' in Africa, and improve postoperative survival.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Biccard, MBChB; PhD, Principal Investigator — UCT
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Biccard BM, Madiba TE, Kluyts HL, Munlemvo DM, Madzimbamuto FD, Basenero A, Gordon CS, Youssouf C, Rakotoarison SR, Gobin V, Samateh AL, Sani CM, Omigbodun AO, Amanor-Boadu SD, Tumukunde JT, Esterhuizen TM, Manach YL, Forget P, Elkhogia AM, Mehyaoui RM, Zoumeno E, Ndayisaba G, Ndasi H, Ndonga AKN, Ngumi ZWW, Patel UP, Ashebir DZ, Antwi-Kusi AAK, Mbwele B, Sama HD, Elfiky M, Fawzy MA, Pearse RM; African Surgical Outcomes Study (ASOS) investigators. Perioperative patient outcomes in the African Surgical Outcomes Study: a 7-day prospective observational cohort study. Lancet. 2018 Apr 21;391(10130):1589-1598. doi: 10.1016/S0140-6736(18)30001-1. Epub 2018 Jan 3. PMID 29306587
- [Result] ASOS-2 Investigators. Enhanced postoperative surveillance versus standard of care to reduce mortality among adult surgical patients in Africa (ASOS-2): a cluster-randomised controlled trial. Lancet Glob Health. 2021 Oct;9(10):e1391-e1401. doi: 10.1016/S2214-109X(21)00291-6. Epub 2021 Aug 19. PMID 34418380
- [Result] O'Cathain A, Croot L, Duncan E, Rousseau N, Sworn K, Turner KM, Yardley L, Hoddinott P. Guidance on how to develop complex interventions to improve health and healthcare. BMJ Open. 2019 Aug 15;9(8):e029954. doi: 10.1136/bmjopen-2019-029954. PMID 31420394
- [Result] Johnston M, Arora S, King D, Stroman L, Darzi A. Escalation of care and failure to rescue: a multicenter, multiprofessional qualitative study. Surgery. 2014 Jun;155(6):989-94. doi: 10.1016/j.surg.2014.01.016. Epub 2014 Feb 7. PMID 24768480
- [Result] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Result] Damschroder LJ, Reardon CM, Widerquist MAO, Lowery J. The updated Consolidated Framework for Implementation Research based on user feedback. Implement Sci. 2022 Oct 29;17(1):75. doi: 10.1186/s13012-022-01245-0. PMID 36309746
- [Result] Baker T, Schell CO, Lugazia E, Blixt J, Mulungu M, Castegren M, Eriksen J, Konrad D. Vital Signs Directed Therapy: Improving Care in an Intensive Care Unit in a Low-Income Country. PLoS One. 2015 Dec 22;10(12):e0144801. doi: 10.1371/journal.pone.0144801. eCollection 2015. PMID 26693728

DOCUMENTS (2):
  • Study Protocol (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT06997328/Prot_000.pdf
  • Statistical Analysis Plan (2026-01-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT06997328/SAP_001.pdf